CLINICAL TRIAL: NCT04255784
Title: A Randomized Sham-Controlled Trial of High-Dosage Accelerated Intermittent Theta Burst rTMS in Major Depression
Brief Title: High Dose Accelerated iTBS for Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: University Health Network, Toronto (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Daniel Blumberger, Medical Head and Co-Director, Temerty Centre for Therapeutic Brain Intervention, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 109-2019
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder
Keywords: depression; transcranial magnetic stimulation; treatment resistance; theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active iTBS (Experimental): Administered 8 times daily at approximately 50 minutes intervals (between session end and start) for 5 days. Each session will deliver 1800 pulses of active iTBS (bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz, with a duty cycle of 2 seconds on, 8 seconds off, over 60 cycles / ~10 minutes) at a target intensity of 110% of the subject's resting motor threshold.
  Interventions: Device: Active iTBS
- Sham iTBS (Sham Comparator): Administered 8 times daily at approximately 50 minutes intervals (between session end and start) for 5 days, using a sham coil that reproduces auditory and tactile sensations of stimulation and has an identical external appearance. Each session will deliver 1800 pulses of sham iTBS (bursts of 3 pulses at 50 Hz, bursts repeated at 5 Hz, with a duty cycle of 2 seconds on, 8 seconds off, over 60 cycles / ~10 minutes) at a target intensity of 110% of the subject's resting motor threshold.
  Interventions: Device: Sham iTBS

INTERVENTIONS:
Device: Active iTBS — Fluid-Cooled B70 A/P Coil with either Magventure X100 or R30
  Arms: Active iTBS
Device: Sham iTBS — Fluid-Cooled B70 A/P Coil with either Magventure X100 or R30
  Arms: Sham iTBS

SUMMARY:
This trial will compare active intermittent theta burst stimulation (iTBS) rTMS in an accelerated treatment schedule (8 treatment sessions per day for 5 days) to a placebo control. Depression symptom severity will be measured before, during, at end of treatment, 1-week post and 4-weeks post treatment.

DETAILED DESCRIPTION:
Those participants who do not meet the response criterion (50% improvement from baseline on the HRDS-17) at the 4-week follow-up will be offered a second course of treatment, regardless of whether they were in the active or the sham treatment group. The blind will be maintained and no further assessment contributing to the primary or secondary outcomes will occur after the 4-week time point. A different operator will administer the open-label second course of treatment to ensure blinding of operators. The second course of treatment will apply active rTMS using low-frequency (1 Hz) stimulation to the right DLPFC for 600 pulses (10 minutes), 8x daily at 50 minutes (between session and end and start) intervals for 5 days. All those completing the second course of treatment will undergo the same set of clinical assessments during and after the course of treatment on the same schedule as the first course of treatment. The final 4-week follow up assessment from the first course of treatment will serve as the baseline for those that go on to receive the second open label treatment course.

ELIGIBILITY:
Inclusion Criteria:

1. are outpatients
2. are voluntary and competent to consent to treatment
3. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of MDD, single or recurrent
4. are between the ages of 18 and 65
5. have failed to achieve a clinical response to an adequate dose of an antidepressant based on an Antidepressant Treatment History Form (ATHF) score for that antidepressant trial of > 3 in the current episode OR have been unable to tolerate at least 2 separate trials of antidepressants of inadequate dose and duration (ATHF score of 1 or 2 on those 2 separate antidepressants)
6. have a score > 18 on the HRSD-17 item
7. have had no increase or initiation of any psychotropic medication in the 4 weeks prior to screening
8. able to adhere to the treatment schedule
9. Pass the TMS adult safety screening (TASS) questionnaire
10. have normal thyroid functioning based on pre-study blood work.

Exclusion Criteria:

1. have a Mini-International Neuropsychiatric Interview (MINI) confirmed diagnosis of substance dependence or abuse within the last 3 months
2. have a concomitant major unstable medical illness, cardiac pacemaker or implanted medication pump
3. have active suicidal intent
4. are pregnant
5. have a lifetime Mini-International Neuropsychiatric Interview (MINI) diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms
6. have a MINI diagnosis of obsessive compulsive disorder, post-traumatic stress disorder (current or within the last year), anxiety disorder (generalized anxiety disorder, social anxiety disorder, panic disorder), or dysthymia, that is assessed by a study investigator to be primary and causing greater impairment than MDD
7. have a diagnosis of any personality disorder, and assessed by a study investigator to be primary and causing greater impairment than MDD
8. have failed a course of ECT in the current episode or previous episode
9. have received rTMS for any previous indication due to the potential compromise of subject blinding
10. have any significant neurological disorder or insult including, but not limited to: any condition likely to be associated with increased intracranial pressure, space occupying brain lesion, any history of seizure except those therapeutically induced by ECT or a febrile seizure of infancy, cerebral aneurysm, Parkinson's disease, Huntington's chorea, multiple sclerosis, significant head trauma with loss of consciousness for greater than 5 minutes
11. have an intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
12. if participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the study
13. clinically significant laboratory abnormality, in the opinion of the one of the principal investigators or study physicians
14. currently take more than lorazepam 2 mg daily (or equivalent) or any dose of an anticonvulsant due to the potential to limit rTMS efficacy
15. non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Change on the 17-item Hamilton Rating Scale for Depression (HRSD-17) | After 5 treatment days
  ITT

SECONDARY OUTCOMES:
Change on the 17-item Hamilton Rating Scale for Depression (HRSD-17) | one week and four weeks post treatment
  ITT
Proportion of participants achieving response (50% reduction in HRSD-17) and remission (HRSD-17 <8) | After 5 treatment days and at 1-week and 4 weeks post-treatment
  ITT
Change on the Beck Depression Inventory-II (BDI-II) | After 5 treatment days and at 1-week and 4 weeks post-treatment
  ITT
Change on the Generalized Anxiety Disorder 7-Item (GAD-7) | After 5 treatment days and at 1-week and 4 weeks post-treatment
  ITT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Blumberger, MD, Principal Investigator — CAMH
Locations (2):
- Canada (2):
  - University of British Columbia, Vancouver, British Columbia
  - CAMH, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodman MS, Vila-Rodriguez F, Barwick M, Burke MJ, Downar J, Hunter J, Kaster TS, Knyahnytska Y, Kurdyak P, Maunder R, Thorpe K, Trevizol AP, Voineskos D, Zhang W, Blumberger DM. A randomized sham-controlled trial of high-dosage accelerated intermittent theta burst rTMS in major depression: study protocol. BMC Psychiatry. 2024 Jan 8;24(1):28. doi: 10.1186/s12888-023-05470-9. PMID 38191370